CLINICAL TRIAL: NCT02209259
Title: The Effect of Questionnaire Content on Measures of Pain Intensity, Magnitude of Disability, and Symptoms of Depression in Patients With Arm Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000666
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Arm Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group 1 (Experimental): The first intervention group will be comprised of patients who will complete PROMIS Upper Extremity Function, pain intensity, PROMIS depression, and the Positive affect negative affect scale (PANAS) after completing the standard PCS.
  Interventions: Other: PROMIS Upper Extremity Function; Other: Pain intensity; Other: PROMIS depression; Other: Positive affect negative affect scale (PANAS); Other: standard PCS
- Intervention Group 2 (Experimental): The second intervention group will be comprised of patients who will complete PROMIS Upper Extremity Function, pain intensity, PROMIS depression, and the Positive affect negative affect scale (PANAS) after completing a positively-adjusted version of the PCS.
  Interventions: Other: PROMIS Upper Extremity Function; Other: Pain intensity; Other: PROMIS depression; Other: Positive affect negative affect scale (PANAS); Other: positively-adjusted version of the PCS
- Control (Experimental): The third group (the control arm) will complete PROMIS Upper Extremity Function, pain intensity, PROMIS depression, and the Positive affect negative affect scale (PANAS).
  Interventions: Other: PROMIS Upper Extremity Function; Other: Pain intensity; Other: PROMIS depression; Other: Positive affect negative affect scale (PANAS)

INTERVENTIONS:
Other: PROMIS Upper Extremity Function
Other: Pain intensity
Other: PROMIS depression
Other: Positive affect negative affect scale (PANAS)
Other: standard PCS
  Arms: Intervention Group 1
Other: positively-adjusted version of the PCS
  Arms: Intervention Group 2

SUMMARY:
The investigators plan a prospective randomized study to see whether negative questions affect measures of mood, pain, or disability. A total of 175 patients will participate at Massachusetts General Hospital.

DETAILED DESCRIPTION:
Patient mood, pain intensity, and magnitude of disability can be measured using questionnaires. The Pain Catastrophizing Scale (PCS) was developed to measure the extent to which the ineffective coping strategy of catastrophic thinking impacts pain experience. It is currently one of the most widely used measures of catastrophic thinking related to pain. The PCS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced 13 thoughts or feelings when experiencing pain. The questions in the PCS are negatively phrased, e.g. "it's terrible and I think it's never going to get any better."

The effect by which exposure to a stimulus influences a response to a later response is called "priming." Priming is the process of activating particular representations or associations in memory just before carrying out an action or task. Priming affects all aspects of human behavior. For example, syntactic priming is the tendency to use syntactic structures that parallel the structures of sentences we have heard recently: a speaker who has just heard a sentence in passive voice is subsequently more likely to use a passive construction himself.

Priming apparently also has affective dimensions. Zajonc performed an experiment where he showed a list of Chinese characters to his test subjects. He subsequently showed the subjects a list of Chinese words and asked them which words they "liked the best." The words containing characters presented in the first list were evaluated more positively. The negative questions in the PCS may prime patients to be more negative in subsequent questionnaires.

Our group has performed multiple studies on the use of certain words, phrases, and concepts in hand and upper extremity surgery. Bossen et al showed that positive or negative wording of MRI reports influences patients' emotional response, satisfaction, and understanding. We are interested in looking at the possibility that certain questionnaires can affect other questionnaires via a priming effect.

We propose a three-arm single blind, randomized (1:1:1) controlled trial to assess whether negative questions of the PCS affect measures of mood, pain, or disability.

Aim:

The aim of this study is to assess whether the negative questions in the PCS affect measures of mood, pain, or disability.

Primary null hypothesis:

There is no difference in Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Function between patients who complete the standard PCS, patients who complete the positively adjusted PCS, and patients who do not complete the PCS.

Secondary null hypothesis:

There is no difference in pain intensity, PROMIS depression, and (Positive Affect Negative Affect Scale) PANAS scores between patients who complete the standard PCS, patients who complete the positively adjusted PCS, and patient who do not complete the PCS.

ELIGIBILITY:
Inclusion Criteria:

* All new and follow-up patients presenting to the Orthopaedic Hand and Upper Extremity Service
* English fluency and literacy

Exclusion Criteria:

* pregnant women
* Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sullivan M J L, Bishop S, Pivik J. The Pain Catastrophizing Scale: Development andvalidation. Psychol Assess 1995, 7: 524-532.
- [Background] Zajonc, R.B. Mere exposure: A gateway to the subliminal. Current Directions in Psychological Science 2001, 10 (6): 224-228.
- [Background] Bossen JK, Hageman MG, King JD, Ring DC. Does rewording MRI reports improve patient understanding and emotional response to a clinical report? Clin Orthop Relat Res. 2013 Nov;471(11):3637-44. doi: 10.1007/s11999-013-3100-x. Epub 2013 Jun 13. PMID 23761176
- [Derived] Claessen FM, Mellema JJ, Stoop N, Lubberts B, Ring D, Poolman RW. Influence of Priming on Patient-Reported Outcome Measures: A Randomized Controlled Trial. Psychosomatics. 2016 Jan-Feb;57(1):47-56. doi: 10.1016/j.psym.2015.09.005. Epub 2015 Oct 1. PMID 26683347

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard PCS: The first intervention group will be comprised of patients who will complete the standard PCS.
- Positively-adjusted PCS: The second intervention group will be comprised of patients who will complete a positively-adjusted version of the PCS.
- Control: The third group (the control arm) will not complete the PCS.
Period: Overall Study
Arm/Group | Standard PCS | Positively-adjusted PCS | Control
Started | 56 | 56 | 56
Completed | 56 | 56 | 56
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PCS | Positively-adjusted PCS | Control | Total
Number analyzed (Participants) | 56 | 56 | 56 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16) | 51 (18) | 56 (15) | 52 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 28 | 89
  Male | 29 | 22 | 28 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 47 | 46 | 50 | 143
  More than one race | 2 | 6 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 56 | 168

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity
Description: A computerized assessment of upper extremity physical function measured at enrollment. The average T score of the U.S. population is 50, so the T score reported compares the study population to the U.S. population, where a T score greater than 50 is better than the average and a T score less than 50 is worse than the average.
Time Frame: 1day
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard PCS | Positively-adjusted PCS | Control
Number analyzed (Participants) | 56 | 56 | 56
T-score | 39 (9.8) | 43 (8.1) | 41 (11)

2. Secondary Outcome: Pain Intensity
Description: 10 point pain scale, where 0 is no pain and 10 is the most pain
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard PCS | Positively-adjusted PCS | Control
Number analyzed (Participants) | 56 | 56 | 56
units on a scale | 3.5 (3.0) | 3.5 (2.9) | 3.3 (2.9)

3. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Depression
Description: A computerized assessment of depression measured at enrollment. The average T score of the U.S. population is 50, so the T score reported compares the study population to the U.S. population, where a T score greater than 50 is worse than the average and a T score less than 50 is better than the average.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard PCS | Positively-adjusted PCS | Control
Number analyzed (Participants) | 56 | 56 | 56
T-score | 47 (8.4) | 48 (7.9) | 48 (8.5)

ADVERSE EVENTS:
Arm/Group | Standard PCS | Positively-adjusted PCS | Control
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes